CLINICAL TRIAL: NCT00575900
Title: Comparison Between Low Carbohydrate Low Fat, Low Carbohydrate High Fat and Balanced Low Fat Diets in the Treatment of Obesity in Adolescents- a Randomized Controlled Trail.
Brief Title: Low Carbohydrates in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Prof. Moshe Phillip, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc003187ctil; Low carbohydrate diets
Record Dates: First submitted 2007-12-16; First posted 2007-12-18 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Obesity
Keywords: Adolescent obesity,; low carbohydrate diets; metabolic risk factors; BMI
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Low carbohydrate and low fat.
  Interventions: Behavioral: dietary intervention
- 2 (Experimental): Low carbohydrate fat rich diet
  Interventions: Behavioral: dietary intervention
- 3 (Active Comparator): A balanced low fat diet
  Interventions: Behavioral: dietary intervention

INTERVENTIONS:
Behavioral: dietary intervention — 12 weeks of dietary intervention

SUMMARY:
A three arms open,randomized interventional study in order to compare the impact of low carbohydrate diets with different protein and fat ratios versus a standard balanced diet on BMI and metabolic parameters in obese adolescents.

55 obese adolescents (12-18y, BMI > 95th percentile) were randomly allocated to one of three 12-weeks diet regimens: low-carbohydrate low-fat, low-carbohydrate high-fat or balanced low-fat diet, followed by 9-months follow-up. Weight, Height, waist circumference, lipid profile, glucose, insulin, liver enzymes, renal functions, C-reactive protein, leptin, ghrelin and resting energy expenditure were measured in the morning after over-night fast at baseline, during the 12-weeks of intervention and after 9-months of follow-up.

DETAILED DESCRIPTION:
A three arms open,randomized interventional study in order to compare the impact of low carbohydrate diets with different protein and fat ratios versus a standard balanced diet on BMI and metabolic parameters in obese adolescents.

Study design:

The study included 12 weeks of intervention followed by 9 months of follow up, between March 2005 to February 2006. Participants were randomly allocated to one of three diet groups.

Group 1: Low carbohydrate, low fat, protein rich diet containing 1200 kcal a day, 60-gr carbohydrates (20%), 40-gr fat (30%), 150-gr protein (50%).

Group 2: Low carbohydrate fat rich diet containing 1200 kcal a day, 60-gr carbohydrates (20%), 80-gr fat (60%), 60-gr protein (20%).

Group 3: A balanced low fat diet containing 1200 kcal a day, 150 - 180-gr carbohydrates (50 - 60%), 40-gr fat (30%), 60-gr protein (20%).

All participant received menus and detailed instruction according to their group.

During the intervention participant attended weekly sessions with a dietitian and a psychologist and a tests and measures scheduled for each time point were performed (see Measures section). In some sessions the participants were requested to fill-out self reports food dairies. All received general recommendations to exercise physical activity.

At the end of the intervention period (12th week), all participants were given instruction for a balanced maintenance diet for the following year.

measures: Anthropometric assessment (weight,height, waist circumference) included baseline and weekly measurement during the 12- week intervention, and thereafter every three months for 9-months of follow-up. Body composition was evaluated at baseline and after the 12- week intervention, after overnight fasting by bioimpedance analysis (BIA). Resting energy expenditure (REE) was assessed at baseline and after the 12- week intervention, in the morning after overnight fasting by means of indirect calorimetry. Urine was collected every week during the intervention period for assay of ketone and protein level. Fasting blood tests were preformed at baseline, weeks 7 and 12, and at the end of the follow-up to measure the following parameters: total cholesterol, Low Density Lipoprotein (LDL), HDL cholesterol, triglycerides, glucose, insulin, blood urea nitrogen, creatinine, total protein, liver enzymes (AST, ALT, GGT ),renal functions (urea, creatinine, electrolytes, uric acid), electrolyte level, Insulin like growth factor (IGF1), haemoglobin, C-reactive protein (CRP), TSH, free T4, iron, vitamin B12, folic acid ,leptin ,and ghrelin.

ELIGIBILITY:
Inclusion Criteria:

1. aged 12 to 18
2. body mass index (BMI) values greater than the 95th percentile for age and gender according to the growth charts of the Center for Disease Control and Prevention.

Exclusion Criteria:

1.Patients with a chronic disease (such as diabetes, renal, heart or liver diseases, thyroid function disorder, or diagnosed psychological disorder). 2.Patients receiving weight-loss-inducing medication.

3.Subjects who had participated in another weight loss-study or slimming diet within two months prior to the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2005-03; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
BMI, BMI-SDS, Body fat percentage, waist circumference | At baseline visit, end of 12 weeks of intervention and every three months after during the 9 months follow-up

SECONDARY OUTCOMES:
Blood metabolic profile, CRP, Ghrelin and Leptin levels, Resting energy expenditure, Psychological parameters | At baseline, after 12 weeks of intervention and after 9 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Rabin Medical Center
Locations (1):
- Schnider children medical center, Petah Tikva, I, Israel